CLINICAL TRIAL: NCT06383897
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and the Impact of Food on Pharmacokinetics of HS-10398 in Healthy Participants, and a Clinical Trial to Assess the Pharmacokinetic Characteristics of HS-10398 in Participants With Kidney Dysfunction
Brief Title: Phase 1 Study in Healthy Participants and Participants With Kidney Dysfunction
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10398-101
Record Dates: First submitted 2023-06-20; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: HS-10398; Phase 1; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort1：HS-10398 (Experimental): SAD： HS-10398 capsule
  Interventions: Drug: HS-10398
- Cohort2：HS-10398 Placebo (Placebo Comparator): SAD：HS-10398 capsule placebo
  Interventions: Drug: HS-10398 Placebo
- Cohort3：HS-10398 (Experimental): MAD： HS-10398 capsule
  Interventions: Drug: HS-10398
- Cohort4：HS-10398 Placebo (Placebo Comparator): MAD：HS-10398 capsule placebo
  Interventions: Drug: HS-10398 Placebo
- Cohort5：HS-10398 (Experimental): HS-10398 capsule will be administered orally once on Day 1 in Participants With Kidney Dysfunction
  Interventions: Drug: HS-10398

INTERVENTIONS:
Drug: HS-10398 — SAD：HS-10398 capsule (5 predefined dose cohorts ) will be administered orally once on Day 1 MAD：HS-10398 capsule (5 predefined dose cohorts ) will be administered orally once or twice from Day 1 to Day 14 IRF：HS-10398 capsule will be administered orally once on Day 1 in Participants With Kidney Dysfunction
  Arms: Cohort1：HS-10398; Cohort3：HS-10398; Cohort5：HS-10398
Drug: HS-10398 Placebo — SAD：HS-10398 capsule placebo (5 predefined dose cohorts ) will be administered orally once on Day 1 MAD：HS-10398 capsule placebo (5 predefined dose cohorts ) will be administered orally once or twice from Day 1 to Day 14
  Arms: Cohort2：HS-10398 Placebo; Cohort4：HS-10398 Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics, and the impact of food on pharmacokinetics of oral HS-10398 in Chinese healthy participants, and a clinical trial to assess the pharmacokinetic characteristics of oral HS-10398 in Chinese participants with kidney dysfunction

DETAILED DESCRIPTION:
This is a phase 1, first-in-human, randomized, double-blind, placebo-controlled, dose-escalation clinical trial. The primary objective is to evaluate the safety, tolerability, and pharmacokinetic characteristics of single and multiple oral doses of HS-10398 in Chinese healthy participants. The secondary objective is to assess the impact of food on the pharmacokinetics of single oral doses of HS-10398 in Chinese healthy participants, as well as to evaluate the pharmacokinetic characteristics of oral HS-10398 in Chinese participants with kidney dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged from 18 to 64 years
* Subjects need to fully understand the research content and process, as well as possible adverse reactions, and voluntarily signed Informed Consent Form
* Males' weight should be ≥ 50kg, and females' weight should be ≥ 45kg. Body mass index (BMI), calculated as weight/height^2 (kg/m^2), should be controlled within the range of 19 to 28, including the critical value
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection is required prior to the start of study treatment. If the patient has not been previously vaccinated, or if a booster is required, vaccine should be given according to local regulations at least 2 weeks prior to first study drug administration
* Participants with Kidney Dysfunction must have met the following additional criteria to be enrolled in this study：Patients with chronic kidney disease (defined as the presence of any markers of kidney damage or an estimated glomerular filtration rate (eGFR) persistently less than 90 mL/min/1.73m² for more than 3 months), and with an estimated glomerular filtration rate (eGFR) at screening and baseline assessments (with a minimum interval of 3 days between screening and baseline assessments) meeting the criteria of 60≤eGFR<90 mL/min/1.73m².

Exclusion Criteria:

* Has a history of chronic or serious disease from neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, metabolic endocrine system, skin disease, blood system, immune system or tumor
* Has taken any drugs, including prescription drugs, over-the-counter drugs, herbal preparations, some health products or inhibitor/inducer of CYP3A4/5 or CYP2C8 or any medications that inhibit P-glycoprotein transporters., within 2 weeks (or 5 half-lives) before screening and throughout the study period
* Has clinically significant ECG abnormalities, such as QT interval corrected according to Fridericia formula(QTcF), >450 ms (males), >470 ms (females)
* Has participated in another clinical trial involving drugs or medical devices within the month prior to screening and received investigational drugs or used medical devices, or within 5 half-lives of the investigational drugs from another trial at the time of screening, whichever is longer
* Unable to abstain from smoking and alcohol.
* History of drug dependence or substance abuse

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From screening to day 15
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Serious adverse events (SAEs) | From screening to day 15
  The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | up to 216 hours after dosing
  Cmax will be obtained following administration of a single oral dose of HS-10398
Time to reach maximum plasma concentration (Tmax) | up to 216 hours after dosing
  Tmax will be obtained following administration of a single oral dose of HS-10398
Elimination Halflife (T1/2) | up to 216 hours after dosing
  Elimination Halflife (T1/2) is the time measured for the concentration to decrease by one half which will be obtained following administration of a single oral dose of HS-10398
Apparent clearance（CL/F） | up to 216 hours after dosing
  CL/F will be obtained following administration of a single oral dose of HS-10398
Apparent Volume of Distribution（Vd/F） | up to 216 hours after dosing
  Vd/F will be obtained following administration of a single oral dose of HS-10398

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, China